CLINICAL TRIAL: NCT03397550
Title: The Relationship Between Salt Restriction and Taste Sensitivity in Patients With Chronic Kidney Disease
Status: Withdrawn | Type: Observational
Why Stopped: feasibility is being questioned
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Dong Jie, Nephrology chief physician, Peking University First Hospital
Other Study IDs: pekingUFH-cn
Record Dates: First submitted 2017-12-13; First posted 2018-01-12 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Renal Insufficiency, Chronic; Chronic Kidney Diseases
Keywords: taste threshold; salt restriction
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: salt restriction education — Salt intake target：<5g/d Method：the standard salt restriction education will be lasting for 10-15 minutes by oral explanation at baseline.

SUMMARY:
The compliance of salt restriction in patients with CKD may be associated with taste sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* stage 3-5 CKD patients
* clinical stable

Exclusion Criteria:

* renal replacement therapy
* cancer
* systemic infection
* Alzheimer's disease
* acute cardiovascular events, active hepatitis
* all other study-obstructive conditions

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: stage 3-5 CKD patients
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-06-18 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
ratings of taste sensitivity assessed by the ISO method of investigating sensitivity of taste（ISO 3972:1991） | up to 12 weeks after intervention
  Taste sensitivity is measured by five taste solutions（salty、sour、bitter、sweet、umami). Every taste solution contains 8 different concentration. Detection , recognition and difference thresholds will be measured .Their definitions are as bellow.
  Detection threshold：minimum value of sensory stimulus needed to give rise to a sensation. The sensation need not be identified.
  Recognition threshold：minimum value of a sensory stimulus permitting identification of the sensation perceived.
  Difference threshold：value of the smallest perceptible difference in the physical intensity of a stimulus.

CONTACTS AND LOCATIONS:
Overall Officials: Jie Dong, Study Director — Peking Universiy First Hospital
Locations (1):
- Peking University First Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Lynch KE, Lynch R, Curhan GC, Brunelli SM. Altered taste perception and nutritional status among hemodialysis patients. J Ren Nutr. 2013 Jul;23(4):288-295.e1. doi: 10.1053/j.jrn.2012.08.009. Epub 2012 Oct 6. PMID 23046735
- [Result] Kusaba T, Mori Y, Masami O, Hiroko N, Adachi T, Sugishita C, Sonomura K, Kimura T, Kishimoto N, Nakagawa H, Okigaki M, Hatta T, Matsubara H. Sodium restriction improves the gustatory threshold for salty taste in patients with chronic kidney disease. Kidney Int. 2009 Sep;76(6):638-43. doi: 10.1038/ki.2009.214. Epub 2009 Jun 10. PMID 19516246
- [Result] Middleton RA, Allman-Farinelli MA. Taste sensitivity is altered in patients with chronic renal failure receiving continuous ambulatory peritoneal dialysis. J Nutr. 1999 Jan;129(1):122-5. doi: 10.1093/jn/129.1.122. PMID 9915887
- [Result] McMahon EJ, Campbell KL, Bauer JD. Taste perception in kidney disease and relationship to dietary sodium intake. Appetite. 2014 Dec;83:236-241. doi: 10.1016/j.appet.2014.08.036. Epub 2014 Sep 2. PMID 25192896